CLINICAL TRIAL: NCT07370753
Title: Early Application of Continuous Renal Replacement Therapy as Adjunctive Support in Pediatric Septic Shock: A Prospective Observational Study
Brief Title: Early Continuous Renal Replacement Therapy for Pediatric Septic Shock
Status: Active, not recruiting | Type: Observational
Sponsor: National Children's Hospital, Vietnam (Other)
Responsible Party: Principal Investigator, Phuc Huu Phan, Principle Investigator, National Children's Hospital, Vietnam
Other Study IDs: IRB-VN01037/IRB00011976/FWA000; DT.007/24 (Other Grant/Funding Number: Vietnam Ministry of Health)
Record Dates: First submitted 2026-01-01; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Sepsis-induced Multiple Organ Dysfunction Syndrome; Septic Shock
Keywords: pediatric sepsis; septic shock; multiple organ dysfunction syndrome; cytokines
MeSH Terms: conditions — Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Septic shock is a major cause of morbidity and mortality in critically ill children. Continuous renal replacement therapy (CRRT) is increasingly used as adjunctive support in pediatric septic shock to improve hemodynamic stability, modulate inflammatory responses, and correct metabolic disturbances. However, evidence regarding optimal indications, timing, and clinical outcomes of early CRRT use in children remains limited.

This prospective observational study aims to evaluate associations between early CRRT use and changes in hemodynamics, organ dysfunction, inflammatory cytokine levels, and short-term clinical outcomes in pediatric patients with septic shock admitted to pediatric intensive care units

DETAILED DESCRIPTION:
This is a prospective observational cohort study conducted in pediatric intensive care units (PICUs). Children diagnosed with septic shock who receive early continuous renal replacement therapy (CRRT) as part of routine clinical care will be consecutively enrolled.

Baseline assessments will be performed prior to CRRT initiation and include clinical status, hemodynamic parameters, echocardiographic indices, laboratory markers, and inflammatory cytokine levels. Follow-up assessments will be conducted at predefined time points after CRRT initiation.

CRRT initiation, modality, and management will follow institutional protocols and treating physician judgment. No randomization or intervention assignment is performed. Patients will be followed during PICU stay and up to Day 28 after PICU admission

ELIGIBILITY:
Inclusion Criteria:

* Age from 1 month to <18 years
* Diagnosis of septic shock according to Phoenix Sepsis Criteria, defined as:

  * Phoenix Sepsis Score ≥ 2, and
  * Presence of circulatory dysfunction
* Fulfillment of at least one of the following:

  * Acute kidney injury KDIGO stage 2 or higher
  * Requirement for vasoactive support with Vasoactive-Inotropic Score (VIS) ≥ 50
* Admission to a Pediatric Intensive Care Unit (PICU)
* Written informed consent obtained from parent(s) or legal guardian(s)

Exclusion Criteria:

* Expected survival <24 hours at time of screening

  o End-stage organ failure, including: End-stage renal disease requiring chronic dialysis or eGFR <15 mL/min/1.73 m²
  * End-stage liver disease
  * End-stage heart failure
* Known immunosuppression, including HIV infection or primary immunodeficiency disorders
* Emergency indications for CRRT unrelated to septic shock (e.g., severe hyperkalemia, severe dysnatremia, symptomatic uremia, or fluid overload >10%)
* PICU length of stay <24 hours
* CRRT duration <6 hours

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with septic shock admitted to the PICU and receiving early continuous renal replacement therapy as part of routine clinical care
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-03-18 (Estimated)

PRIMARY OUTCOMES:
Time to shock reversal | From initiation of CRRT until first documented shock reversal, assessed up to 7 days after CRRT initiation during PICU stay
  Shock reversal is defined as sustained improvement in hemodynamic stability, including reduction of vasoactive support, normalization of age-adjusted heart rate and blood pressure, arterial lactate <2 mmol/L, and central venous oxygen saturation (ScvO₂) between 70-75%.
Change in Pediatric Sequential Organ Failure Assessment (pSOFA) Score | Baseline, 24 hours, 48 hours, 72 hours, Day 5, and Day 7 after CRRT initiation
  Change in organ dysfunction severity assessed using the Pediatric Sequential Organ Failure Assessment (pSOFA) score (range: 0-24), with higher scores indicating more severe organ dysfunction

SECONDARY OUTCOMES:
Change in mean arterial pressure (MAP) | Time Frame: Baseline, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours after CRRT initiation
  Change in mean arterial pressure measured after initiation of continuous renal replacement therapy (CRRT), unit of measurement is mmHg
Change in serum cytokine levels | Baseline, 12 hours, 24 hours, and 48 hours after CRRT initiation
  Change in serum cytokine concentrations, including tumor necrosis factor alpha (TNF-α), interleukin-1 (IL-1), interleukin-6 (IL-6), interleukin-12 (IL-12), interferon gamma (IFN-γ), interleukin-10 (IL-10), transforming growth factor beta (TGF-β), and interleukin-4 (IL-4), measured after initiation of continuous renal replacement therapy (CRRT).
  All cytokines will be measured using the same assay platform and reported in the same unit of concentration. Unit of measurement is pg/ml
Changes in serum lactate concentration | Baseline, 6 hours, 12 hours, 24 hours, 48 hours, and 72 hours after CRRT initiation
  Change in serum lactate concentration measured after initiation of continuous renal replacement therapy (CRRT). Unit of measurement is mmol/L
Mortality outcomes | up to day 28
  All-cause mortality at Day 7 All-cause mortality at Day 28

OTHER OUTCOMES:
ICU resource utilization | up to Day 28
  ICU-free days: calculated as 28 minus ICU length of stay for patients discharged alive before Day 28; assigned 0 for patients who die before Day 28 or remain in ICU on/after Day 28.
  Ventilator-free days: calculated as 28 minus days of invasive mechanical ventilation for patients alive and ventilated <28 days; assigned 0 for patients who die before Day 28 or remain ventilated on/after Day 28.
  Vasopressor-free days: calculated as 28 minus days receiving vasoactive agents for patients alive and requiring vasoactives <28 days; assigned 0 for patients who die before Day 28 or remain on vasoactives on/after Day 28. Discontinuation requires ≥12 hours without vasoactive support

CONTACTS AND LOCATIONS:
Locations (1):
- Vietnam National Children's Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT07370753/Prot_SAP_000.pdf